CLINICAL TRIAL: NCT01623128
Title: Prenatal Education Video Study
Acronym: PEVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Virginia Department of Health (Other Government)
Responsible Party: Principal Investigator, Ann Kellams, MD, Prinicpal Investigaor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 14812
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Breastfeeding
Keywords: Breastfeeding initiation; Breastfeeding duration; WIC; Video education; Breastfeeding rates
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Breastfeeding video (Experimental): Participants randomized to this arm view the intervention video - Injoy Videos Better Breastfeeding video.
  Interventions: Behavioral: Prenatal video
- Sham video (Placebo Comparator): Participants randomized to this arm view the sham video Injoy Videos Your Healthy Pregnancy: Prenatal Nutrition and Exercise video.
  Interventions: Behavioral: Prenatal video

INTERVENTIONS:
Behavioral: Prenatal video — Participants are randomized to view either the intervention video or a sham video.
  Other Names: Injoy videos

SUMMARY:
A randomized, controlled trial will be conducted during which pregnant women will be randomized to receive the intervention - viewing a prenatal education video about how to breastfeed an infant - or the sham intervention - viewing a prenatal education video about maternal nutrition and physical activity during pregnancy. Participants will be interviewed via telephone at one, three, and six months post-partum to determine how they feed their infants at each of these time frames.

DETAILED DESCRIPTION:
Research assistants will screen potential candidates at the University of Virginia Health System and Virginia Commonwealth University Primary Care Center and approach potential participants during a standard clinic visit. The charts of the day's patients will be screened prior to approaching women to invite them to enroll in the study.

Following administration of the enrollment questionnaire, the patient will be randomized to the intervention or sham intervention arm of the study. The research assistant will open the study packet with the corresponding study identification number containing the intervention assignment. The research assistant will then load the assigned video into the DVD player and ask the patient to view the video. The participants will be blinded to which video is the true intervention.

Following delivery, research assistants will abstract the medical records of the woman and infant. Data regarding complications for both the mother and baby will be recorded and the length of stay for mother and baby as well as information about the way in which the baby was fed during the hospital stay.

Participants will be administered a one-month follow-up questionnaire by telephone. Follow-up questionnaires will be administered by research staff that did not enroll the participant such that the research assistant administering the telephone questionnaire will be blinded to the patient's assigned intervention group. The three-month questionnaire will be administered by telephone in the same fashion as the one-month. The six-month questionnaire will be administered by telephone. This questionnaire will conclude the study. A current address will be obtained at this time, and a children's book will be mailed to the participant thanking her for completing the study. For subjects lost to follow-up, we will contact the baby's pediatrician to retrieve the information on the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Receiving prenatal care at the Primary Care Center, University Physicians for Women at Northridge, the University of Virginia Teen Health Center
* WIC-eligible 185% Federal poverty Enrolled in Medicaid, TANF, food stamps
* Pregnant, 24 - 41 weeks gestation
* Singleton gestation
* Access to a telephone
* Plan to deliver at UVa
* Primary language is English or Spanish

Exclusion Criteria:

* Multiple gestation
* Known contraindication to breastfeeding Illicit drug use HIV + Recipient of chemotherapy
* Primary language other than English or Spanish

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 522 (Actual)
Dates: Start 2010-03; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Breastfeeding | 6 months post-partum
  To determine the effect of the intervention on the initiation, duration, and exclusivity of breastfeeding among low-income, WIC-eligible women.

SECONDARY OUTCOMES:
Infant feeding practices for women that deliver prior to 35 weeks gestation | Six months post-partum
  To determine the effect of the intervention on infant feeding practices immediately postpartum among women who deliver their babies prior to 35 weeks of gestation.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Kellams, MD, Principal Investigator — University of Virginia School of Medicine
Locations (2):
- United States (2):
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia